CLINICAL TRIAL: NCT03770130
Title: Evaluation of the Impact of Dexmedetomidine on Allograft Function Recovery and Survival Following Liver Transplantation: A Randomised Control Trial
Brief Title: Dexmedetomidine and Liver Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS-OLT Trial
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Dexmedetomidine, Liver Transplantation, Allograft Function, Survival
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine treatment group (Experimental): Anaesthesia will be maintained with sevoflurane inhalation, of which the concentration will be adjusted to maintain the BIS value between 40 and 60. Muscle relaxation will be maintained with rocuronium or cisatracurium. Analgesia will be maintained with remifentanil (administered via continuous infusion), sufentanil (administered via continuous infusion or intermittent injection), or fentanyl (administered via intermittent injection). In addition to this, patients will receive an initial loading dose of dexmedetomidine of 1μg/kg over 10 min after the induction of anaesthesia followed by a continuous infusion of 0.5μg/kg/h until the end of surgery.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Anaesthesia will be maintained with sevoflurane inhalation, of which the concentration will be adjusted to maintain the BIS value between 40 and 60. Muscle relaxation will be maintained with rocuronium or cisatracurium. Analgesia will be maintained with remifentanil (administered via continuous infusion), sufentanil (administered via continuous infusion or intermittent injection), or fentanyl (administered via intermittent injection). In addition to this, patients will receive an equal volume initial loading dose of 0.9% saline over 10 min after the induction of anaesthesia followed by an equal volume continuous infusion until the end of surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine, a selective α2-adrenoceptor agonist which is widely used as an adjuvant to general anaesthesia
  Arms: Dexmedetomidine treatment group
Drug: Saline — Saline, a kind of crystalloid widely used in clinical treatment
  Arms: Control group

SUMMARY:
1.1. Background 1.1.1. Perioperative ischaemia/reperfusion (I/R) injury during liver transplantation is strongly associated with early allograft dysfunction, graft loss, and mortality.

1.1.2. Hepatic I/R injury also causes remote damage to other organs including the renal and pulmonary systems.

1.1.3. Dexmedetomidine, a selective α2-adrenoceptor agonist which is widely used as an adjuvant to general anaesthesia, has been widely shown in preclinical studies to provide organoprotection by ameliorating the effects of I/R injury in a range of tissues (including the liver). However, prospective clinical evidence of any potential benefits in improving outcomes in liver transplantation is lacking.

1.2. Objectives 1.2.1. To investigate the hypothesis that perioperative treatment with dexmedetomidine reduces the incidence of early allograft dysfunction and primary graft non-function in deceased donor liver transplantation.

1.2.2. The impact of dexmedetomidine on postoperative renal and pulmonary function will also be examined.

1.3. Study Design This is a prospective, single-centre, randomised, parallel-group study.

1.4. Setting Departments of Anesthesiology, Renji Hosptial, Shanghai Jiao Tong University School of Medicine, Shanghai, 200127, China.

1.5. Patients 200 patients (18-65 years) scheduled to undergo liver transplantation under general anaesthesia.

1.6 Intervention 1.6.1. For the patients in the treatment group, a loading dose of dexmedetomidine will be given after induction of anaesthesia (1μg/kg over 10 min) followed by a continuous infusion (0.5μg/kg /h) until the end of surgery.

1.6.2. For patients in the placebo group, an equal volume loading dose of 0.9% saline will be given after the induction of anaesthesia followed by an equal volume continuous infusion until the end of surgery.

1.6.3. All other supplements, e.g. opioids, sedatives and muscle relaxant, will be identical in the both arms and administered according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Scheduled to undergo allogenic liver transplant(DCD/DBD) surgery under general anaesthesia
3. Patients should meet the UCSF criteria
4. Agree to participate and give written informed consent

Exclusion Criteria:

1. Severe renal dysfunction (undergoing renal replacement therapy before surgery)
2. Severe pulmonary dysfunction (including pneumonia, atelectasis, pleural effusion, acute lung injury or ARDS)
3. Severe circulatory instability (severe coronary artery disease, unstable angina, left ventricular ejection fraction < 30%, sick sinus syndrome, severe sinus bradycardia [< 50 bpm], second-degree or greater atrioventricular block)
4. Known allergy or intolerance to trial medication
5. Refusal to participate in the study
6. Participation in other clinical trials within 30 days prior to randomisation.
7. Retransplantation
8. Multiple organ transplantation
9. Other reasons that are considered unsuitable for study participation by the responsible surgeon or anaesthetist (reasons must be documented in the case report form [CRF])

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of early allograft dysfunction (EAD) following surgery | 7 days
  Defined according to Olthoff's criteria published in 2010: (1) bilirubin ≥ 10mg/dL on day 7; or (2) INR > 1.6 on day 7; or (3) AST/ ALT > 2000IU/L within first 7 days.

SECONDARY OUTCOMES:
Incidence of postoperative acute kidney injury (AKI) during the postoperative day 1-7 | 7 days
  Defined by Kidney Disease: Improving Global Outcomes (KDIGO) criteria published in 2012: (1) Increase in serum creatinine by ≥ 0.3mg/dL within 48 hours; or (2) increase in serum creatinine to 1.5 times baseline or more within past 7 days; or (3) urine output < 0.5mL/kg/h for 6 hours.
Incidence of acute respiratory distress syndrome (ARDS) during the postoperative day 1-7 | 7 days
  Defined according to Berlin modification of the American European Consensus Committee (AECC) definitions published in 2012: (1) Acute onset (within one week of known insult); and (2) bilateral opacities on CXR (not explained by effusions, nodules, or collapse); and (3) respiratory failure not fully explained by cardiac failure or fluid overload; and (4) Severity graded by PaO2/ FIO2 ratio with PEEP 5cmH2O i. Mild 300 ≥ PaO2/ FIO2 > 200; ii. Moderate 200 ≥ PaO2/ FIO2 > 100; iii. Severe 100 ≥ PaO2/ FIO2.
Incidence of graft failure and retransplantation rate during 3 year follow up period. | 3 years
All cause mortality in the 3 year follow-up period. | 3 years
Incidence of primary graft non-function (PNF) | 30 days
  Defined as graft loss, retransplantation, or patient death due to graft non-function in first 30 days (excluding non-function secondary to hepatic artery thrombosis, biliary complications, or recurrent hepatic disease).

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Yang L, Zhu L, Qi B, Zhang Y, Ni C, Zhang Y, Shi X, Xia Q, Masters J, Ma D, Yu W. Dexmedetomidine use during orthotopic liver transplantation surgery on early allograft dysfunction: a randomized controlled trial. Int J Surg. 2024 Sep 1;110(9):5518-5526. doi: 10.1097/JS9.0000000000001669. PMID 38768468
- [Derived] Ni C, Masters J, Zhu L, Yu W, Jiao Y, Yang Y, Cui C, Yin S, Yang L, Qi B, Ma D. Study design of the DAS-OLT trial: a randomized controlled trial to evaluate the impact of dexmedetomidine on early allograft dysfunction following liver transplantation. Trials. 2020 Jun 26;21(1):582. doi: 10.1186/s13063-020-04497-7. PMID 32591004